CLINICAL TRIAL: NCT06783491
Title: Efficacy of the Use of Neoadjuvant With/Without Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Colon Cancer: A Phase III Multi-arm, Randomized and Controlled Clinical Trial (FOXHIPECT4)
Brief Title: Efficacy of the Use of Neoadjuvant With/Without Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Colon Cancer
Acronym: FOXHIPECT4
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other); Spanish Association of Surgeons (AEC) (Other); Sociedad Española de Oncología Quirúrgica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCO-FOX-2025-01; 2025-520471-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Colorectal Cancer
Keywords: colorectal cancer; hyperthermic intraperitoneal chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mitomycin; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Cytoreduction Surgical Procedures

STUDY DESIGN:
Intervention Model Description: controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FOLFOX+SURGERY+HIPEC (Experimental): FOLFOX x6 (12 weeks) followed by cytoreductive surgery + HIPEC (mitomycin 30mg/m2 for 60 min) followed by FOLFOX x6 (12 weeks).
  Interventions: Drug: Mitomycin (MM); Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin); Procedure: Cytoreductive surgery
- FOLFOX+SURGERY (Experimental): FOLFOX x6 (12 weeks) followed by cytoreductive surgery followed by FOLFOX x6 (12 weeks).
  Interventions: Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin); Procedure: Cytoreductive surgery
- cytoreductive surgery + standard care (Active Comparator): cytoreductive surgery followed by standard care (adjuvant therapy according to local protocol). Cytoreductive surgery will be defined as complete tumour resection including oncologic colectomy and adjacent structures with suspicious of infiltration to achieve a R0, bilateral oophorectomy is recommended in post-menopausal women.
  Interventions: Procedure: Cytoreductive surgery

INTERVENTIONS:
Drug: Mitomycin (MM) — Mitomycin 30mg/m2/4 litres of perfusion liquid (dextrose 1.5%). Single intraoperative dose.
  Arms: FOLFOX+SURGERY+HIPEC
Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin) — FOLFOX6 consists in oxaliplatin 85 mg/m2 iv. on day 1, 5FU 400 mg/m2 iv. in bolus followed by 2400 mg/m2 in a continuous infusion for 46 hours. Leucovorin: 400mg/m2 folinic acid (racemid dl) in a continuous infusion for 2 hours. Repeat every 2 weeks. Haematological recovery to ANC >1.5x109/L and platelets >75x109/L should be ensured prior to Day 1 of each 14-day cycle.
  Arms: FOLFOX+SURGERY; FOLFOX+SURGERY+HIPEC
Procedure: Cytoreductive surgery — Cytoreductive surgery will be defined as complete tumour resection including oncologic colectomy and adjacent structures with suspicious of infiltration to achieve a R0, bilateral oophorectomy is recommended in post-menopausal women

SUMMARY:
The main objective of this randomized and controlled trial is to determine whether the use of a proactive strategy, systemic neoadjuvant treatment (FOLFOX) with or without hyperthermic intraperitoneal chemoterapy (HIPEC) with mitomycin C followed by postoperative systemic adjuvant treatment, increases disease-free survival at 36 months in patients with locally advanced colon cancer compared to standard treatment. Therefore, a phase III, randomized, academic, multicenter, controlled trial will be conducted. Patients with locally advanced colon adenocarcinoma (cT4, cT3 with invasion >5mm) Nx and no metastases will be included. Control group (n=361) will receive standard treatment (surgery and adjuvant chemotherapy FOLFOX x 12 based); Experimental group 1 (n=361) = Neoadjuvant chemotherapy (FOLFOX x6) + surgery (associating HIPEC) and FOLFOX x 6; Experimental group 2 (n=361): Neoadjuvant chemotherapy (FOLFOX x6) + surgery and FOLFOX x 6. Randomization will be 1:1:1, stratified and centralized. The primary outcome will be disease-free survival at 36 months. Secondary outcomes will be tumor regression rate, ctDNA negativization, peritoneal relapse rate at 36 months, pattern of relapse, toxicity, morbidity and overall survival. Considering the results obtained with these two independent strategies (FOLFOX and HIPEC), a new trial is justified in order to provide strong evidence for this proactive treatment. The aim is to combine both to obtain a better benefit, which opens the direct possibility of increasing the current percentage of disease-free survival. The results of this study will have important scientific and social impact, since is aimed at improving the outcomes of one subpopulation of patients with locally advanced colon cancer whose current treatment, is not enough to avoid the recurrence of disease.

DETAILED DESCRIPTION:
he MAIN HYPOTHESIS of this trial is that the combination of systemic neoadjuvant chemotherapy with hyperthermic intraperitoneal chemotherapy (HIPEC) will have a synergistic effect in preventing disease recurrence (at all levels) in patients with locally advanced colorectal cancer.

Therefore, the GENERAL OBJECTIVE of this study is to determine whether the use of proactive systemic neoadjuvant treatment (FOLFOX) with or without HIPEC with mitomycin C followed by post-surgical systemic adjuvant treatment increases disease-free survival at 36 months in patients with locally advanced colon cancer compared to standard treatment. To achieve this general goal, we will implement the following specific objectives (SO):

SO1: To determine the efficacy of neoadjuvant systemic treatment with or without HIPEC association disease-free survival (DFS) at 36 months.

SO2: To conduct a stratified analysis by factors including tumor location (right/left), definitive pathologic stage II/III (high risk), sex and age.

SO3: To evaluate tumor regression after neoadjuvant treatment using the Dworak tumor regression scale (grade 0-no regression to grade 5-total response).

SO4: To evaluate the R0 surgery rate in the different treatment groups.

SO5: To compare the circulating tumor DNA (ctDNA) detected after surgery in both, experimental and control groups and analyze its impact in survival according to its detection.

SO6: To evaluate the morbidity and toxicity in the different treatment groups.

SO7: To determine the efficacy of neoadjuvant systemic treatment with or without HIPEC association in peritoneal (local or diffuse) recurrence-free survival (PFS) at 36 months.

SO8: To evaluate the effect of neoadjuvant therapy associated with HIPEC compared to neoadjuvant treatment on the pattern of disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged ≥18 years and ≤75 years (patients between 70-75 years old will be discussed in committee).
* Adenocarcinoma of the colon, sigmoid colon and rectum-sigmoid junction that is cT4a/b according to the American Joint Committee on Cancer (AJCC) TNM eight edition. Pre-treatment diagnosis by imaging test (CT scan or MRI). High-risk cT3 with invasion into surrounding fat greater than 5mm may be included.
* Nodal extension: cN0, the presence of cN1/2 according to AJCC TNM 8th edition is allowed as long as they can be resected. Pre-treatment diagnosis by imaging test (CT scan or MRI).
* Metastatic extension: cM0. Patients with cM1 are not allowed to be included.
* ECOG 0-1.
* Microsatellite stability (pMMR).
* Informed consent duty completed.

Exclusion Criteria:

* Presence of metastases (M1). If liver or peritoneal metastases are present at the time of surgery, the patient will be excluded from the study and treated according to the new stage.
* Presence of un-resectability criteria in the pretreatment work-up, un-resectability will be discussed in MDT with expert oncologic surgeons.
* Presence of microsatellite instability (dMMR).
* Presence of deficit of DPD.
* Urgent intervention due to obstruction or perforation if the primary tumour is removed. Bridge interventions such as transit shunts without removal of the primary tumour or percutaneous drainage of collections prior to neoadjuvant treatment or scheduled surgery will be accepted.
* Extraperitoneal rectal cancer (medium-low) (avoiding alterations due to neoadjuvant radiotherapy).
* Coexistence of another relevant malignant neoplastic disease (synchronous colon and rectum-sigmoid tumours are accepted as long as the stage is equal or lower than the treated tumour), it will be discussed in steering committee.
* Severely impaired hepatic, renal or cardiovascular function.
* Intolerance to treatment.
* Gestational or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1083 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival absolute | 36 months after treatment.
  Absolute disease-free survival in months. The event will be defined by patient death from any cause or tumour recurrence
Disease-free survival probability | 36 months after treatment.
  Tumour disease-free survival at 3 years of follow-up (%). The event will be defined by patient death from any cause or tumour recurrence up to 36 months after treatment.

SECONDARY OUTCOMES:
Absolute Overall survival | 36 months after treatment.
  The event will be defined by patient death from any cause
Probability overall survival | 36 months after treatment.
  Probability of survival at 3 years. The event will be defined by patient death from any cause up to 36 months after treatment
Tumour regression | 12 weeks after treatment
  Tumour regression grade (Dworak's scale)
ctDNA rate | 36 months after treatment.
  Negative rate of ctDNA after treatment and association of detected levels with tumour recurrence and survival.
Absolute Disease-free survival in subgroups | 36 months after treatment.
  Absolute disease-free survival in months in the following subgroups: pT4a/b/pT3b, pN+, pathologic stage II/III, right/left colon cancer mutated RAS/RAF, positive/negative ctDNA. The event will be defined by patient death from any cause or tumour recurrence
Disease-free survival probability in subgroups | 36 months after treatment.
  Tumour disease-free survival at 3 years of follow-up (%) in the following subgroups: pT4a/b/pT3b, pN+, pathologic stage II/III, right/left colon cancer mutated RAS/RAF, positive/negative ctDNA. The event will be defined by patient death from any cause or tumour recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Arjona Sánchez, MD., Ph.D., Principal Investigator — MAIMONIDES BIOMEDICAL RESEARCH INSTITUTE
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided